CLINICAL TRIAL: NCT04994418
Title: The Impact of Sodium and Fructose on Blood Pressure and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, William Farquhar, Professor, University of Delaware
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1617405-2
Record Dates: First submitted 2021-04-16; First posted 2021-08-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Blood Pressure; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1. Recommended sodium and low fructose diet (Experimental): 7 day consumption of low fructose drink (20g) and recommended sodium (2300mg) from whole food while consuming placebo from pills
  Interventions: Dietary Supplement: High sodium and low fructose diet; Dietary Supplement: High sodium and high fructose diet
- Arm 2. High sodium and low fructose diet (Experimental): 7 day consumption of low fructose drink (20g) and recommended sodium (2300 mg) from whole food while consuming high sodium from pills (3400 mg)
  Interventions: Dietary Supplement: Recommended sodium and low fructose diet; Dietary Supplement: High sodium and high fructose diet
- Arm 3. High sodium and high fructose diet (Experimental): 7 day consumption of high fructose drink (200g) and recommended sodium (2300 mg)from whole food while consuming high sodium pills from pills (3400 mg)
  Interventions: Dietary Supplement: Recommended sodium and low fructose diet; Dietary Supplement: High sodium and low fructose diet

INTERVENTIONS:
Dietary Supplement: Recommended sodium and low fructose diet — Upon completion of a 7 day dietary intervention of consuming the daily recommended sodium and low fructose contents we will investigate changes in ambulatory blood pressure, urinary sodium excretion, heart rate variability, secretion of inflammatory cytokines, and reactive oxygen species.
  Arms: Arm 2. High sodium and low fructose diet; Arm 3. High sodium and high fructose diet
Dietary Supplement: High sodium and low fructose diet — Upon completion of a 7 day dietary intervention of consuming the daily high sodium and low fructose contents we will investigate changes in ambulatory blood pressure, urinary sodium excretion, heart rate variability, secretion of inflammatory cytokines, and reactive oxygen species.
  Arms: Arm 1. Recommended sodium and low fructose diet; Arm 3. High sodium and high fructose diet
Dietary Supplement: High sodium and high fructose diet — Upon completion of a 7 day dietary intervention of consuming the high sodium and high fructose contents we will investigate changes in ambulatory blood pressure, urinary sodium excretion, heart rate variability, secretion of inflammatory cytokines, and reactive oxygen species.
  Arms: Arm 1. Recommended sodium and low fructose diet; Arm 2. High sodium and low fructose diet

SUMMARY:
The goal of this study is to determine the impact of dietary sodium and fructose on blood pressure and inflammation in young healthy adults.

DETAILED DESCRIPTION:
Excess dietary salt is associated with an increased risk of cardiovascular diseases. Some healthy adults have been determined to be more sensitive to dietary salt than others, which can result in a 10% or more increase of blood pressure. The mechanisms underlying salt sensitivity of blood pressure are not fully understood. Previous research has suggested excess intake of added sugars, especially fructose, can increase salt sensitivity of blood pressure. Chronic elevated consumption of salt and fructose independently have been shown to have damaging effects on the body, however, the combination of both salt and fructose has not been fully studied in humans. The purpose of this research study is to determine if increased dietary fructose consumption will stimulate salt-sensitive hypertension and induce proinflammatory cytokines through activation of the immune system. Understanding how the body regulates blood pressure during times of elevated salt and fructose is important for determining cardiovascular risk in a population with normal blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* normal blood pressure
* males, females, minorities

Exclusion Criteria:

* high blood pressure
* body mass index (BMI) of > 30 kg/m2
* smokers or nicotine users
* pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
24-hour Blood Pressure | Day 7 of diet intervention
  Systolic blood pressure over 24 hours (mmHg)
Inflammatory cytokines | Day 7 of diet intervention
  ELISA assay detecting Interleukin-6 and tumor necrosis factor-alpha

CONTACTS AND LOCATIONS:
Overall Officials: Ronald K McMillan, M.S, Principal Investigator — University of Delaware; William B Farquhar, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Undecided